CLINICAL TRIAL: NCT05130671
Title: Treatment Benefits of Flavonoids Quercetin and Curcumin Supplements for Mild Symptoms of COVID-19
Brief Title: Nutritional Supplementation of Flavonoids Quercetin and Curcumin for Early Mild Symptoms of COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, somia iqtadar, Associate Professor of Medicine, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 785/RC/KEMU/25.10.2021
Record Dates: First submitted 2021-11-21; First posted 2021-11-23 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care; Therapies, Investigational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): This arm will receive the standard of care as per the hospital guidelines.
  Interventions: Drug: Standard of care
- Investigational treatment (Experimental): This arm will receive combination of nutritional supplements quercetin and curcumin as add-on to the standard of care.
  Interventions: Drug: Standard of care; Dietary Supplement: Investigational treatment

INTERVENTIONS:
Drug: Standard of care — Standard of care treatment as per the hospital guidelines
Dietary Supplement: Investigational treatment — Combination of quercetin and curcumin as add-on to the standard of care
  Arms: Investigational treatment

SUMMARY:
The purpose of this study is to investigate the therapeutic benefits of flavonoids nutritional supplements quercetin and curcumin for early mild symptoms of COVID-19.

DETAILED DESCRIPTION:
Flavonoids nutritional supplements quercetin and curcumin have demonstrated strong antioxidant, broad-spectrum anti-viral and anti-inflammatory properties including against the respiratory tract infections. They are widely used to boost the immunity against infections and keeping healthy life-style. Results from recent published studies have shown positive results for quercetin and curcumin in patients with COVID-19.

In the present study the investigators aim to study the combined beneficial effects of quercetin and curcumin in addition to standard of care for managing early mild symptoms of COVID-19 in community-based patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older, of either gender
* Patients must be tested positive for SARS-CoV-2 by RT-PCR
* Patients must exhibit typical symptoms of COVID-19 disease at screening such as fever, fatigue, a dry and contagious cough, loss of appetite, body aches, shortness of breath, mucus or phlegm, sore throat, headache, chills, sometimes withshaking, loss of smell or taste, congestion or runny nose, nausea, or vomiting, diarrhea, muscular pain etc.
* Patients must be in the early stage of COVID-19 disease who do not require hospitalization at the time of screening
* Patients must be under the care of a Physician for diagnosis of COVID-19
* Patients who have signed informed consent

Exclusion Criteria:

* Patients with proven hypersensitivity or allergic reaction to quercetin or curcumin
* Patients with known chronic kidney disease with estimated creatinine clearance < 50 mL/minute or need for dialysis
* Patients who are severely hypotensive defined as needing hemodynamic pressors to maintain blood pressure
* Patients taking anticoagulant/antiplatelet drugs such as Coumarine, Heparine, Aspirin, Clopidrogel, dalteparin, enoxaparin, ticlopidine and warparin.
* Patients with gallstone obstruction
* Hypothyroid suppering patients
* Patients with moderate or severe thrombocytopenia (platelet count <100 ×10⁹/L);
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Testing negative for SARS-CoV-2 by Reverse Transcription Polymerase Chain Reaction (RT-PCR) | Day 7
  Testing of naso-pharyngeal swab for COVID-19
COVID-19 symptoms improvement | Day 7
  Improvement of the typical symptoms associated with COVID-19 infection

SECONDARY OUTCOMES:
Improvement in CRP level | Day 7
  Improvement in the CRP levels
Improvement in D-dimers level | Day 7
  Improvement in D-dimers level
Improvement in LDH levels | Day 7
  Improvement in LDH levels
Improvement in ferritin levels | Day 7
  Improvement in Ferritin levels
Improvement in full blood count (CBC) | Day 7
  Improvement in CBC levels

CONTACTS AND LOCATIONS:
Locations (1):
- King Edward Medical University Teaching Hospital, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Derived] Khan A, Iqtadar S, Mumtaz SU, Heinrich M, Pascual-Figal DA, Livingstone S, Abaidullah S. Oral Co-Supplementation of Curcumin, Quercetin, and Vitamin D3 as an Adjuvant Therapy for Mild to Moderate Symptoms of COVID-19-Results From a Pilot Open-Label, Randomized Controlled Trial. Front Pharmacol. 2022 Jun 7;13:898062. doi: 10.3389/fphar.2022.898062. eCollection 2022. PMID 35747751